CLINICAL TRIAL: NCT05969509
Title: Investigation of the Effect of Progressive Relaxation Exercises on Pain and Bowel Movements in Patients Undergoing Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Şuheda Zorer, principal investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AtaturkU-SBF-SZ-01
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: two groups consisting of experimental and control groups performed cholecystectomy.
Who Masked: Outcomes Assessor
Masking Description: the cholecystectomy group will be given exercise sessions and the result evaluations will be performed by a researcher who is blind to the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the group that performed relaxation exercises (Experimental): patients' postoperative pain and bowel movements will be evaluated by applying relaxation exercise intermittently
  Interventions: Other: progressive relaxation exercise
- the group that did not do relaxation exercises (No Intervention): patients' postoperative pain and bowel movements will be evaluated

INTERVENTIONS:
Other: progressive relaxation exercise — applying progressive relaxation exercise to the experimental group after postoperative cholecystectomy and observing the experimental-control groups
  Arms: the group that performed relaxation exercises

SUMMARY:
The goal of this clinical trial is to compare in health conditions. The main questions it aims to answer are:

Does progressive relaxation exercises reduce pain in patients undergoing laparoscopic cholecystectomy? Does progressive relaxation exercises increase bowel movements in patients undergoing laparoscopic cholecystectomy?

DETAILED DESCRIPTION:
The purpose of our experimentally randomized controlled study, which researchers conducted in order to study the effect of progressive relaxation exercises on pain and bowel movements in patients undergoing laparoscopic cholecystectomy, is to reduce pain by intermittent application of progressive relaxation exercises to patients after surgery and to study the effect of exercise on bowel movements at an early stage.

after the necessary permissions have been obtained july- september dates, Van Yüzüncü yıl university Dursun Odabaş medical center, in the general surgery clinic , patients who agree to participate in the study and meet the sample selection criteria will be included in the study. Patient presentation form, bowel movement monitoring form and Visual Analog Scale (VAS) Pain Form will be used in the collection of research data.

ELIGIBILITY:
Inclusion Criteria:

* Who experienced laparoscopic cholecystectomy surgery as planned for the first time
* Who volunteered to participate in the research
* 18 years and over
* Whose mental state is healthy
* Without vision, hearing and speech problems
* Patients who know Turkish were included in the study.

Exclusion Criteria:

* Who have previously practiced progressive relaxation exercises
* Someone with communication problems
* Health problems that prevent the practice of progressive relaxation exercises (Epilepsy, bipolar disorder, schizophrenia, fever, infection, etc. ) is
* Patients who were not willing to participate in the study were not included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Pain Form | examination between 1-2 days until Decontamination from surgery
  it is a scale with two ends named differently on the vertical or horizontal line with a length of 10 cm (0=no pain, 10=the most severe pain). Marking the point corresponding to the intensity of pain felt by the patient on this line
bowel movement monitoring form | examination between 1-2 days until Decontamination from surgery
  It is the form in which the intestinal sounds, gas extraction and defecation sounds of the patients are monitored by the researcher.

CONTACTS AND LOCATIONS:
Overall Officials: şuheda zorer, Principal Investigator — van yüzüncü yıl university dursun odabaş medical center
Locations (1):
- Van Yüzüncü Yıl University Dursun Odabaş Medical Center, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zorer Yilmaz S, Gurcayir D. The Effect of Progressive Relaxation Exercises on Pain and Bowel Movements in Patients Undergoing Laparoscopic Cholecystectomy: A Randomized Controlled Trial. Asian Nurs Res (Korean Soc Nurs Sci). 2025 Oct;19(4):410-416. doi: 10.1016/j.anr.2025.08.004. Epub 2025 Sep 18. PMID 40975381